CLINICAL TRIAL: NCT02426294
Title: A Phase IV, Multicenter, Randomized, Active Comparator Controlled Study of the Addition of Pioglitazone Compared With Glimepiride in Subjects With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Metformin and Alogliptin
Brief Title: Comparison of Pioglitazone Versus Glimepiride in Type 2 Diabetes Inadequately Controlled With Metformin Plus Alogliptin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, In Ju Kim, Department of Internal Medicine, Pusan National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALO-IIT-013
Record Dates: First submitted 2015-03-07; First posted 2015-04-24 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pioglitazone (Experimental): Pioglitazone is a Pioglitazone hydrochloride, and white circle-shaped tablet. It is administered once-daily with 15mg, with or without meals. The once-daily administration begins with 15mg, and if need increase, researchers can increase up to 30mg at week 12.
  Interventions: Drug: Pioglitazone
- Glimepiride (Active Comparator): The generic name of Glimepiride is Glimepiride, and it is a green snowman-shaped tablet. The once-daily administration begins with 2mg, and if need increase, researchers can increase up to 4mg at week 12.
  Interventions: Drug: Glimepiride

INTERVENTIONS:
Drug: Pioglitazone
  Other Names: Actos
  Arms: Pioglitazone
Drug: Glimepiride
  Other Names: Amaryl
  Arms: Glimepiride

SUMMARY:
The purpose of this study is to compare the treatment effect at week 26 between the two groups, sulfonylurea (SU, glimepiride) administration and thiazolidinedione (TZD, Pioglitazone) administration, as the third-order drug among patients whose treatment is not sufficient after the combined administration of Metformin and Alogliptin.

DETAILED DESCRIPTION:
1. Background Complications of diabetes could cause death from stroke and myocardial infarction, and it is the chronic disease that leads to foot amputation, blindness and renal failure. According to the data of Statistics Korea, the prevalence rate of diabetes for people over 30 years old (standardization) has gradually increased from 8.6% in 2001 to 9.7% in 2010. Although diabetes is not the direct cause of death or disability, it is becoming a significant health problem across the world as it is a major illness causing complications.

   Diabetic complications are very common; the patients of end-stage renal failure with diabetes were 56.7% and patients who begin renal replacement therapy with diabetes were 70.5% in 2003. The prevalence rate of eye problems including cataract, retinopathies and glaucoma in diabetic patients is 1.9 times higher than that in non-diabetic patients. In addition, it is estimated that the incidence rate of acute stroke, which is a complication of the great vessels of diabetic patients, is also 5.2 times higher than that of the general population. As diabetes could cause various complications and be dangerous, the regulation of blood glucose level is essential in order to prevent these complications.

   According to the Korea National Health & Nutrition Examination Survey in 2008~2010, the rate of patients with well-controlled glycated hemoglobin of below 6.5% among diabetic patients over 30 years old is only 25%. Thus, many studies are being conducted to lower the glycated hemoglobin by administering various line drugs, alone or in combination, because the regulation of blood glucose is difficult for many diabetic patients.

   When the regulation of blood glucose ends in failure with a single dose of a drug, the combination treatment is recommended. Metformin is mainly used as the first-order treatment drug, and the second and third drugs, such as dipeptidyl peptidase-4 (DPP-4) inhibitor and sulphonylurea, are recommended to use if the first one is not sufficient.

   DPP-4 inhibitor is a new line of hypoglycemic agent based on incretin. It has statistically significant results for the regulation of glycated hemoglobin compared to existing oral hypoglycemic agents.

   Therefore, many clinicians use Metformin as the first-order drug, and DPP-4 inhibitor as the second-order drug. Alogliptin, which was recently proved to have no side effects of the cardiovascular system, is effective in the regulation of blood glucose as well as the weight control and the prevention of hypoglycemia. Moreover, it is effective when administered alone, and also effective when coadministered with Metformin, Glibenclamide and Pioglitazone. In particular, the reduction degree of glycated hemoglobin was significantly larger when it was administered with Pioglitazone.

   Sulphonylurea, the most well-known hypoglycemic agent, is helpful in the regulation of blood glucose and reduces the occurrence frequency of hypoglycemia when combined with Metformin.
2. Rationale This study examines the related factors of the Pioglitazone group, which is a TZDs line, and the Glimepiride group, which is a sulphonylurea line, as the third-order drugs for patients who are coadministered Metformin and Alogliptin, a DPP-4 inhibitor.
3. Hypothesis When the SU and TZDs drugs administered as third-order drugs in the patients who administered second-order drugs, the treatment effect is different between the two drugs
4. Primary Aim/Objective:

   The primary objective is to compare the mean changes of HbA1c at week 26 between the two groups, SU (glimepiride) administration and TZDs (Pioglitazone) administration, as the third-order drug among patients whose treatment is not sufficient after the combined administration of Metformin and Alogliptin.
5. Primary Endpoint(s):

The mean changes of HbA1c at week 26 from baseline

ELIGIBILITY:
Inclusion Criteria:

* Subjects included in the study are regular type 2 diabetes outpatients of male and female with a level of 7.5%≤HbA1c<10%, despite metformin and alogliptin treatments more than 3months, between 19 and 80 years old.
* Patients had to have a body weight of at least 55 kg and or a body mass index of 22-35 kg/m2

Exclusion Criteria:

* the use of weight-lowering drugs, any investigational blood-glucose or lipid-lowering agent (other than statins or ezetimibe) within the past 3 months
* previous treatment with systemic corticosteroids or a change in dosage of thyroid hormones in the previous 6 weeks
* the use of insulin within the 3 months prior to screening
* allergy or hypersensitivity to target medication or any of its components
* history of type 1 diabetes; acute metabolic complications of diabetes (e.g. ketoacidosis or hyperosmolar state (coma or precoma)) within the preceding 6 months
* haematological disorders
* history of angioedema with angiotensin converting enzyme inhibitors or angiotensin receptor blockers, or treated diabetic gastric paresis
* renal failure, moderate or severe renal impairment (creatinine clearance<50 ㎖/min; or estimated glomerular filtration rate<50 ㎖/min/1.73㎡) before screening
* Serious heart failure or prior history of heart failure(NYHA Class Ⅲ or Ⅳ heart failure.
* impaired hepatic function (defined as elevated serum levels of either alanine aminotransferase, aspartate aminotransferase or alkaline phosphatase 2.5-fold the upper limit of the normal range [ULN] or elevated serum total bilirubin levels 2.5-fold ULN)
* hereditary complications (limited to lactose containing medicines) such as galactose intolerance, deficiency of Lapp lactase, glucose-galactose malabsorption syndrome, etc
* cardiovascular disease, myocardial infarction, or in the previous 6 months; coronary angioplasty, coronary stent placement
* serious cerebrovascular, stroke, transient ischemic attack in the previous 6 months
* laser treatment for proliferative diabetic retinopathy
* history of alcohol or drug abuse in the previous 3 months
* history of all of cancers not in remission for 5 years
* Active bladder cancer
* experience of a major operation
* premenopausal women who were nursing or pregnant were also ineligible for trial participation
* external injury, acute infections, a history/presence of any other severe disease, or severe trauma
* fasting plasma glucose (FPG) level of >239.6mg/dL
* systolic or diastolic blood pressure >160 mmHg or >100 mmHg, respectively
* serum creatinine level of >1.5mg/dL for men or 1.3mg/dL for women
* fasting cholesterol >250mg/dL
* thyroid-stimulating hormone higher than the upper limit of normal
* hemoglobin level is below 12 g/dL for men and below 10 g/dL for women
* fasting triglyceride levels> 5.1 mmol/l (452 mg/dL)

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-12 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Evidence of efficacy of glycemic control indicated by the mean changes of HbA1c (%) at week 26 from baseline | 26 weeks

SECONDARY OUTCOMES:
Evidence of changes of insulin resistance and secretion at week 26 from baseline | 26 weeks
  Homeostatic model assessment model
Evidence of changes of Lipid profile at week 26 from baseline | 26 weeks
  LDL (Low-density lipoprotein) cholesterol, HDL (high-density lipoprotein) cholesterol and triglyceride
Evidence of efficacy of glycemic control indicated by the mean changes of HbA1c (%) at week 12 from baseline | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: In Joo Kim, MD., PhD., Principal Investigator — Pusan National University Hospital
Locations (1):
- Pusan National University Hospital, Busan, South Korea

REFERENCES:
- [Derived] Kim JM, Kim SS, Kim JH, Kim MK, Kim TN, Lee SH, Lee CW, Park JY, Kim ES, Lee KJ, Choi YS, Kim DK, Kim IJ. Efficacy and Safety of Pioglitazone versus Glimepiride after Metformin and Alogliptin Combination Therapy: A Randomized, Open-Label, Multicenter, Parallel-Controlled Study. Diabetes Metab J. 2020 Feb;44(1):67-77. doi: 10.4093/dmj.2018.0274. Epub 2019 Jul 11. PMID 31339011